CLINICAL TRIAL: NCT02269267
Title: The Life After Stopping Tyrosine Kinase Inhibitors Study (The LAST Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: University of Chicago (Other); University of California, San Francisco (Other); University of Utah (Other); Dana-Farber Cancer Institute (Other); Emory University (Other); Barbara Ann Karmanos Cancer Institute (Other); Duke Cancer Institute (Other); Fred Hutchinson Cancer Center (Other); Memorial Sloan Kettering Cancer Center (Other); Weill Medical College of Cornell University (Other); H. Lee Moffitt Cancer Center and Research Institute (Other)
Responsible Party: Principal Investigator, Ehab L Atallah, Professor (Principal Investigator), Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00023447
Record Dates: First submitted 2014-10-08; First posted 2014-10-21 (Estimated); Results first posted 2023-03-01 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Leukemia, Myeloid, Chronic
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate; Dasatinib; nilotinib; bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Discontinuation of TKI medication (Other): Patients with CML on treatment with imatinib, dasatinib, nilotinib, or bosutinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years.
  Interventions: Drug: Imatinib (Stopping their TKI); Drug: Dasatinib (Stopping their TKI); Drug: Nilotinib (Stopping their TKI); Drug: Bosutinib (Stopping their TKI)

INTERVENTIONS:
Drug: Imatinib (Stopping their TKI) — Patients with CML on treatment with imatinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years. Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with PCR testing, though at fewer time points, utilizing online and/or phone questionnaires.
  Other Names: Gleevec
Drug: Dasatinib (Stopping their TKI) — Patients with CML on treatment with dasatinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years. Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with PCR testing, though at fewer time points, utilizing online and/or phone questionnaires.
  Other Names: Sprycel
Drug: Nilotinib (Stopping their TKI) — Patients with CML on treatment with nilotinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years. Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with PCR testing, though at fewer time points, utilizing online and/or phone questionnaires.
  Other Names: Tasigna
Drug: Bosutinib (Stopping their TKI) — Patients with CML on treatment with bosutinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years. Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with PCR testing, though at fewer time points, utilizing online and/or phone questionnaires.
  Other Names: BOSULIF

SUMMARY:
This is a non-randomized, prospective, single-group longitudinal study. The purpose of this study is to improve the decision making process used by physicians and patients when they are considering stopping their Tyrosine Kinase Inhibitor (TKI) medication.

DETAILED DESCRIPTION:
This is a non-randomized, prospective, single-group longitudinal study. The overall objective is to improve decision making for TKI discontinuation in eligible chronic myelogenous leukemia (CML) patients. Patients with CML on treatment with imatinib, dasatinib, nilotinib, or bosutinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years. The study will closely monitor patients using standard real-time Quantitative Polymerase Chain Reaction (RQ-PCR) testing for molecular recurrence, testing them monthly for six months, then every other month until 24 months, and then quarterly until 36 months. Concurrently, the study will assess a wide range of patient-reported outcomes (PROs) before stopping TKIs and after discontinuation in conjunction with Polymerase Chain Reaction (PCR) testing, though at fewer time points, utilizing online and/or phone questionnaires. Patients who have molecular CML recurrence based on RQ-PCR will restart imatinib, dasatinib, nilotinib, or bosutinib and will continue to be monitored for disease status and health status until the end of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 or older at time of study entry
2. Willing and able to give informed consent
3. Diagnosed with CML in chronic phase and have either the b3a2 (e14a2) or b2a2 (e13a2) variants that give rise to the p210 BCR-ABL protein
4. Currently taking imatinib, dasatinib, nilotinib or bosutinib
5. Patient has been on TKI therapy for at least 3 years
6. Documented BCR-ABL <0.01% (>MR4 i.e. >4 log reduction) or undetectable BCR-ABL by PCR for at least 2 years according to the patient's local lab
7. Documented BCR-ABL <0.01% (>MR4 i.e. >4 log reduction) or undetectable BCR-ABL at least 3 times prior to screening according to the patient's local lab
8. Two (2) Screening PCRs have been completed and both results are < 0.01% (>MR4 i.e > 4 log reduction) by central lab
9. Has been on any number of TKIs, but has not been resistant to any TKI (changes made for intolerance are allowed)
10. Patient has been compliant with therapy per treating physician

Exclusion Criteria:

1. Prior hematopoietic stem cell transplantation
2. Poor compliance with taking TKI
3. Unable to comply with lab appointments schedule and PRO assessments
4. Life expectancy less than 36 months
5. Patients who have been resistant to previous TKI therapy are not eligible
6. Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 173 (Actual)
Dates: Start 2014-12-18 (Actual); Primary Completion 2021-04-06 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ehab Atallah, MD, Principal Investigator — Medical College of Wisconsin; Kathryn Flynn, PhD, Principal Investigator — Medical College of Wisconsin
Locations (16):
- United States (16):
  - Helen Diller Family Comprehensive Cancer Center University of California, San Francisco, California
  - Moffit Cancer Center, Tampa, Florida
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - The University of Chicago, Chicago, Illinois
  - The University of Chicago Medicine Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Beth Israel Deaconess Medical Center (Satellite site of Dana Farber), Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute of Wayne State University, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Medical College of Cornell University, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - MD Anderson Cancer Center, Houston, Texas
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - Froedtert Hospital & Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Atallah E, Schiffer CA, Weinfurt KP, Zhang MJ, Radich JP, Oehler VG, Pinilla-Ibarz J, Deininger MWN, Lin L, Larson RA, Mauro MJ, Moore JO, Ritchie EK, Shah NP, Silver RT, Wadleigh M, Cortes J, Thompson J, Guhl J, Horowitz MM, Flynn KE. Design and rationale for the life after stopping tyrosine kinase inhibitors (LAST) study, a prospective, single-group longitudinal study in patients with chronic myeloid leukemia. BMC Cancer. 2018 Apr 2;18(1):359. doi: 10.1186/s12885-018-4273-1. PMID 29609532
- [Result] Atallah E, Schiffer CA, Radich JP, Weinfurt KP, Zhang MJ, Pinilla-Ibarz J, Kota V, Larson RA, Moore JO, Mauro MJ, Deininger MWN, Thompson JE, Oehler VG, Wadleigh M, Shah NP, Ritchie EK, Silver RT, Cortes J, Lin L, Visotcky A, Baim A, Harrell J, Helton B, Horowitz M, Flynn KE. Assessment of Outcomes After Stopping Tyrosine Kinase Inhibitors Among Patients With Chronic Myeloid Leukemia: A Nonrandomized Clinical Trial. JAMA Oncol. 2021 Jan 1;7(1):42-50. doi: 10.1001/jamaoncol.2020.5774. PMID 33180106

RESULTS

PARTICIPANT FLOW:
Groups:
- Discontinuation of TKI Medication: Patients with CML on treatment with imatinib, dasatinib, nilotinib, or bosutinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years.
  Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with polymerase chain reaction (PCR) testing, though at fewer time points, utilizing online and/or phone questionnaires.
Period: Overall Study
Arm/Group | Discontinuation of TKI Medication
Started | 173 (One subject expired prior to achieving an appropriate response for suspension of TKI therapy. Total evaluable subjects = 172 for subsequent analyses.)
Completed | 168
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Groups:
- Discontinuation of TKI Medication: Patients with CML on treatment with imatinib, dasatinib, nilotinib, or bosutinib and are in confirmed deep molecular response will stop their TKI. Confirmed deep (> 4 log reduction) molecular response (>MR4) defined as p210 (bcr-abl) fusion protein (BCR-ABL) < 0.01%, for at least two years.
  Concurrently, the study will assess a wide range of PROs before stopping TKIs and after discontinuation in conjunction with PCR testing, though at fewer time points, utilizing online and/or phone questionnaires.
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 123
  >=65 years | 49
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89
  Male | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 153
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 139
  More than one race | 0
  Unknown or Not Reported | 17
Region of Enrollment [Number; unit: participants]
  United States | 172

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Chronic Myeloid Leukemia (CML) Who Develop Molecular Recurrence After Discontinuing TKIs.
Description: The number of patients who develop molecular recurrence after discontinuing TKIs. This will be reported as the number of new occurrences from the end of the prior time frame.
Time Frame: 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 27, 30, 33, 36 months
Population: One subject expired after the 10th month visit.
Measure: Count of Participants; unit: Participants
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
Participants
  Less or equal to one month | 0
  One month to two months | 4
  Two months to three months | 12
  Three months to four months | 11
  Four months to five months | 7
  Five months to six months | 5
  Six months to eight months | 2
  Eight months to 10 months | 3
  Ten months to 12 months: number analyzed (Participants) | 171
  Ten months to 12 months | 4
  12 months to 14 months: number analyzed (Participants) | 171
  12 months to 14 months | 2
  14 months to 16 months: number analyzed (Participants) | 171
  14 months to 16 months | 2
  16 months to 18 months: number analyzed (Participants) | 171
  16 months to 18 months | 1
  18 months to 20 months: number analyzed (Participants) | 171
  18 months to 20 months | 0
  20 months to 22 months: number analyzed (Participants) | 171
  20 months to 22 months | 0
  22 months to 24 months: number analyzed (Participants) | 171
  22 months to 24 months | 1
  24 months to 27 months: number analyzed (Participants) | 171
  24 months to 27 months | 1
  27 months to 30 months: number analyzed (Participants) | 171
  27 months to 30 months | 2
  30 months to 33 months: number analyzed (Participants) | 171
  30 months to 33 months | 0
  33 months to 36 months: number analyzed (Participants) | 171
  33 months to 36 months | 0
  36 months: number analyzed (Participants) | 171
  36 months | 2

2. Primary Outcome: Patient-reported Health Status Related to Fatigue of Patients at Baseline (Before Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: Patient-reported health status of fatigue using the Patient-Reported Outcomes Measurement Information System (PROMIS) scales. The research team used five questions. The responses are in a Likert -style scale numbered one to five -- 1 (not at all) and 5 (very much). PROMIS scales use a T-score metric for interpretation of results. The mean score for a relevant reference population (United States general population in this case) is 50 and 10 is the standard deviation of that population. T-score range is 20 to 80. Thus, a score of 40 is one standard deviation lower than the reference population mean and a score of 60 is one standard deviation higher than the reference population mean. Higher scores for this scale are indicative of worse symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 52.9 (9.9)

3. Primary Outcome: Patient-reported Health Status Related to Fatigue of Patients at 6 Months (After Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: as for outcome 2
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 50.2 (11.1)

4. Primary Outcome: Patient-reported Health Status Related to Diarrhea of Patients at Baseline (Before Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: Patient-reported health status of diarrhea using the Patient-Reported Outcomes Measurement Information System (PROMIS) scales. There are two unrelated questions. Question no. 1 focuses on loose or watery stool and asks how many days the subject experienced this. O is no days and 4 is six to seven days. Question no. 2 asks if the subject often feels the need to empty the bowel right away. Responses are 0 (never) to 4 (more than once a day). Responses are a Likert -style scale numbered one to five -- 1 (not at all) and 5 (very much). PROMIS scales use a T-score metric interpret results. The mean score for a relevant reference population (United States general population) is 50 and 10 is the standard deviation of the population. T-score range is 20 to 80. A score of 40 is one standard deviation lower than the reference population mean and 60 is one standard deviation higher than the reference population mean. Higher scores indicate worse symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 43.6 (8.3)

5. Primary Outcome: Patient-reported Health Status Related to Diarrhea of Patients at 6 Months (After Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: as for outcome 4
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 40.8 (9.2)

6. Primary Outcome: Patient-reported Health Status Related to Sleep Status of Patients at Baseline (Before Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: Patient-reported health status of sleep using the Patient-Reported Outcomes Measurement Information System (PROMIS) scales. There are four questions. The responses are in a Likert Scale numbered one to five. All questions are regarding the quality of sleep. The answers are one (not at all) to 5 (very much). PROMIS scales use a T-score metric interpret results. The mean score for a relevant reference population (United States general population) is 50 and 10 is the standard deviation of the population. T-score range is 20 to 80. A score of 40 is one standard deviation lower than the reference population mean and 60 is one standard deviation higher than the reference population mean. Higher scores indicate worse symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 49.7 (8.2)

7. Primary Outcome: Patient-reported Health Status Related to Sleep Status of Patients at 6 Months (After Stopping Tyrosine Kinase Inhibitors (TKIs)
Description: as for outcome 6
Time Frame: Six months
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Discontinuation of TKI Medication
Number analyzed (Participants) | 172
T-Score | 48.3 (9.6)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Discontinuation of TKI Medication
All-Cause Mortality (participants affected / at risk) | 5/173
Serious Adverse Events (participants affected / at risk) | 5/173
Other Adverse Events (participants affected / at risk) | 173/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinuation of TKI Medication (N=173)
Suicide attempt (Psychiatric disorders) | 1 (1)
Stroke (Nervous system disorders) | 1 (1)
Death, cause not specified (General disorders) | 2 (2)
Disease progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Discontinuation of TKI Medication (N=173)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Eye "puffiness." bilateral
Eye disorders - Other, specify (Eye disorders) | 1 (1) — Increased difficulty reading
Watering eyes (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 8 (8)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Edema limbs (General disorders) | 3 (3)
Edema limbs (General disorders) | 9 (9)
Fatigue (General disorders) | 20 (20)
Night sweats (General disorders) | 1 (1)
Gout (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pain (General disorders) | 7 (7)
Bladder infection (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 4 (4)
Investigations - Other, specify (Investigations) | 1 (1) — Increased BUN
Investigations - Other, specify (Investigations) | 1 (1) — Ferritin Increased
Platelet count decreased (Investigations) | 2 (2)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1) — Hyperlipidemia
Arthralgia (Musculoskeletal and connective tissue disorders) | 23 (23)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Bone pain (Musculoskeletal and connective tissue disorders) | 6 (6)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 9 (9)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Arthralgia; bilateral shoulders
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Pain (Right Hip, Buttock)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Hamstring Tear
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Right Shoulder Pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle Aches
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Hand Cramping
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Muscle Pain
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Joint Stiffness
Neck pain (Musculoskeletal and connective tissue disorders) | 15 (15)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9)
Concentration impairment (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 5 (5)
Headache (Nervous system disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 6 (6)
Anxiety (Psychiatric disorders) | 3 (3)
Delirium (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 8 (8)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 3 (3)
Nail discoloration (Skin and subcutaneous tissue disorders) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Eczema
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Skin discoloration
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Hair coarsening
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Knot on inner thigh
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Hypersensitivity to right hip and right elbow
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Itching
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) — Rash
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (3)
Hot flashes (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT02269267/Prot_SAP_000.pdf